CLINICAL TRIAL: NCT05169385
Title: Improving Outcomes of Adolescents in Residential Substance Use Treatment Via a Technology-Assisted Parenting Intervention
Brief Title: Parent SMART (Substance Misuse in Adolescents in Residential Treatment)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006002748; R37DA052918 (NIH)
Record Dates: First submitted 2021-12-13; First posted 2021-12-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Substance Use; Adolescent Behavior
Keywords: adolescent; substance use; substance-related disorders
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Effectiveness Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent SMART (Experimental): Parent SMART is a technology-assisted parenting intervention combining an off-the-shelf computer program (Parenting Wisely), up to four telehealth coaching sessions, and access to an app-based networking forum.
  Interventions: Behavioral: Parent SMART
- Treatment as Usual (Active Comparator): The active comparator is defined as residential treatment services as usual.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Parent SMART — Parent SMART experimental intervention
  Arms: Parent SMART
Behavioral: Treatment as Usual — Residential treatment as usual
  Arms: Treatment as Usual

SUMMARY:
Adolescents in residential substance use treatment have serious substance-related problems and poor outcomes following discharge: follow-up studies indicate that 60% of adolescents treated in residential treatment will relapse within the first 90 days. Parenting practices have been established as a critical predictor of adolescents' substance use outcomes and likelihood of relapse following treatments, but parents are notoriously difficult to engage in adolescent substance use treatment. Findings such as these provide strong justification for targeting parents of adolescents in residential substance use treatment via easily accessible interventions.

This study tests the effectiveness of a technology-assisted parenting intervention called Parent SMART (Substance Misuse among Adolescents in Residential Treatment). The intervention combines an off-the-shelf computer program that teaches parenting skills called Parenting Wisely, four telehealth coaching sessions, and a networking forum that allows parents to connect with a clinical expert and with other parents. The investigators will compare adolescents who receive standard residential substance use treatment to adolescents who receive the same treatment plus whose parents receive Parent SMART. Investigators will test the comparative effectiveness of Parent SMART versus residential treatment as usual on parental monitoring and communication, adolescent substance use (i.e., days of substance use and substance-related problems), and substance-related high-risk behaviors (i.e., school-related problems, criminal involvement, externalizing behavior). The investigators will also test whether improvements in parenting partially mediate any observed changes in adolescent substance use and other high-risk behaviors.

DETAILED DESCRIPTION:
Building upon a successful National Institute on Drug Abuse (NIDA)-funded R34, this study evaluates a technology-assisted parenting intervention with evidence of high feasibility and acceptability, as well as preliminary evidence of effectiveness as an adjunct to residential treatment as usual (TAU). Specifically, this study involves a fully powered evaluation of Parent SMART (Substance Misuse among Adolescents in Residential Treatment), which was developed based on extensive formative research with parents, adolescents, and residential treatment staff, and subsequently tested in a NIDA-funded pilot trial.

Parent SMART was intentionally designed with scalability in mind. It consists of an off-the-shelf computer program called Parenting Wisely (PW) that has robust evidence of efficacy in improving parenting skills and reducing youth behavior problems across five clinical trials. Guided by formative research, Parent SMART augments PW with four telehealth coaching sessions and access to a state-of-the-art, mobile networking forum (available via both mobile phone app and web browser), where parents can submit questions to an expert and connect with other parents of adolescents in residential substance use treatment. Parent SMART was piloted at both short (i.e., 6-10 day length of stay) - and long-term (i.e., 30-45 day length of stay) residential facilities: the model was feasible and acceptable in both settings, and effective at improving parental monitoring and communication in both settings. In the short-term setting, Parent SMART was also effective at reducing days of substance use (i.e., days of binge drinking, days of all other drug use) and reducing school problems: the pilot project was underpowered to detect differences at the long-term setting. The current trial is a fully powered evaluation of Parent SMART as an adjunct to residential treatment as usual.

Adolescent-parent dyads (n = 220; 440 participants) will be randomized to receive either residential treatment as usual (TAU) only or Parent SMART + TAU. Those randomized to TAU will be offered the technology-delivered elements of Parent SMART at the 6-month follow-up. Parent SMART telehealth sessions will be delivered by bachelor's and master's level counselors to enhance scalability. Multi-method follow-up assessments (i.e., self-report measures, videotaped interaction task, urine screens) will be conducted 6-, 12-, and 24-weeks post-discharge.

The primary aims of this study is to examine the effectiveness of Parent SMART as an adjunctive treatment, relative to adolescent residential treatment-as-usual on: parenting processes (Primary Aim 1) and adolescent substance use outcomes (Primary Aim 2). A secondary aim is to test the effectiveness of Parent SMART compared to residential treatment-as-usual on adolescent high-risk behaviors. An additional Exploratory Aim will test whether change in parenting processes mediates change in adolescent substance use outcomes.

Pursuit of these aims is significant given the potential to improve the outcomes of adolescents following discharge from residential substance use treatment by offering their parents a novel technology-assisted intervention. Technology-assisted interventions have the potential for marked public health impact by extending the reach, duration, and scalability of evidence-based care.

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* admitted to residential treatment due to concerns about frequency and/or severity of substance use
* report alcohol and/or drug use in the past 90 days
* be discharged to live with primary guardian
* fluent in English or Spanish
* willing and able to participate in a 2 hour interview prior to discharge from residential

Exclusion Criteria for Adolescents:

* does not report alcohol or drug use in the past 90 days
* discharge plan does not include living with primary guardian
* not fluent in English or Spanish
* not willing or able to complete baseline interview

Inclusion Criteria for Parents:

* parent or legal guardian of adolescent aged 12-18 years inclusive, at project start
* adolescent admitted to residential treatment due to concerns about frequency and/or severity of substance use
* will be primary guardian living with adolescent after discharge from residential
* fluent in English or Spanish
* willing and able to complete the baseline assessment prior to the adolescent's discharge
* access to a smartphone that can receive text messages and reliably access the internet

Exclusion Criteria for Parents:

* not legal guardian of adolescent or adolescent not aged between 12-18 years
* adolescent not admitted to residential treatment due to substance use concerns
* will not be living with adolescent after adolescent's discharge from residential
* not fluent in English or Spanish
* not willing or able to complete the baseline assessment prior to the adolescent's discharge
* does not have access to a smartphone that can receive text messages and reliably access the internet

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Monitoring | Baseline to 24 Weeks Post Discharge
  The Parental Monitoring Questionnaire (PMQ), a parent-report and adolescent-report measure, will be used to assess dimensions of parental monitoring. It has three subscales: Child Disclosure, Parent Solicitation, and Parental Control.
Change in Parental Communication | Baseline to 24 Weeks Post Discharge
  The Parent-Adolescent Communication Scale (PCAS), a parent-report and adolescent-report measure, will be used to assess dimensions of parental monitoring. It has two subscales: General Communication and Problems with Communication.
Change in Family Assessment Task Interaction Ratings | Baseline to 24 Weeks Post Discharge
  The Family Assessment Task, a video-taped family problem solving task will be used to provide an in vivo assessment of parenting behavior. Three tasks provide data on monitoring and communication: Limit Setting, Substance Use Norms, and Monitoring and Listening. Tapes will be coded by two raters blind to condition.
Change in Proportion of Days Used Over the Past 90 Days Outside of a Controlled Environment | Baseline to 24 Weeks Post Discharge
  The Global Appraisal of Individual Needs - Core is a well-validated clinical interview used to assess adolescent substance use in a range of settings. Substance consumption information is collected using a calendar format with temporal cues (e.g., holidays) to assist in recall of days when alcohol and other drugs were used. Possible number of days range from 0 to 90. Values are adjusted to reflect the percent of days used outside of controlled environment, with final values ranging from 0 to 100%.
Change in Substance Use Problems | Baseline to 24 Weeks Post Discharge
  The Global Appraisal of Individual Needs - Core is a well-validated clinical interview used to assess adolescent substance use in a range of settings. The Substance-Related Problems Scale provides a count of substance-related problems experienced over the past 90 days. Possible values range from 0 to 11.

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Becker, Ph.D., Principal Investigator — Brown University and Northwestern University
Locations (3):
- United States (3):
  - Rosecrance Health Network, Rockford, Illinois
  - Rosecrance Jackson Centers, Sioux City, Iowa
  - Hazelden Betty Ford, Plymouth, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan for the primary outcomes will be submitted to the Journal of Medical Internet Research Protocols. Additional data (analytic code, participant-level data) can be requested from the Principal Investigator. Analysis files will be constructed from the stored electronic data and will be stripped of identifying information. Specifically, participants will be identified with a numeric identifier that is not related to any element of their personal identifying information. No names, addresses, telephone numbers, fax numbers, email addresses, medical record numbers, etc. will be retained in the de-identified files.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol will be submitted for publication in 2021. Analytic code and participant-level data will be made ready for distribution within 12 months of study completion.
Access Criteria: Data will only be shared with external investigators when a data use agreement (DUA) is executed between Brown University and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data destruction.

REFERENCES:
- [Derived] Patel-Syed Z, Helseth SA, Rosales R, Janssen T, Scott K, Becker SJ. The effects of neighborhood perceptions on response to a technology-assisted parenting intervention for adolescent substance use: protocol of a diversity supplement to parent SMART (Substance Misuse in Adolescents in Residential Treatment). Addict Sci Clin Pract. 2024 Oct 18;19(1):75. doi: 10.1186/s13722-024-00509-y. PMID 39425208
- [Derived] Becker SJ, Helseth SA, Kelly LM, Janssen T, Wolff JC, Spirito A, Wright T. Parent SMART (Substance Misuse in Adolescents in Residential Treatment): Protocol of a Randomized Effectiveness Trial of a Technology-Assisted Parenting Intervention. JMIR Res Protoc. 2022 Feb 28;11(2):e35934. doi: 10.2196/35934. PMID 35225821